CLINICAL TRIAL: NCT03890081
Title: Coping Strategies Questionnaire: Translation, Cultural Adaptation, Reliability and Validity in Turkish-Speaking Subjects With Chronic Musculoskeletal Pain
Brief Title: Reliability and Validity of the Turkish Version of the Coping Strategies Questionnaire
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ugur Sozlu, Research assistant, Gazi University
Other Study IDs: E.70271
Record Dates: First submitted 2019-03-21; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: Coping Strategies Questionnaire; Cross-cultural adaptation; Reliability; Validity
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Translate and culturally adapt the original English version of the Coping Strategies Questionnaire into Turkish

SUMMARY:
Chronic musculoskeletal pain is a major health problem in 35% of the general population in most developed countries. In addition to interventional therapies, the cognitive and behavioral abilities of the patient, are important for the solution of chronic pain. All of these abilities of patients are called coping strategies of pain.

DETAILED DESCRIPTION:
The Coping Strategies Questionnaire (CSQ) is commonly used to measure methods of coping with various forms of chronic pain, including musculoskeletal pain. CSQ aims to evaluate the frequency and success of coping strategies with cognitive and behavioral pain. The validity and reliability of the questionnaire was tested and satisfactory results were obtained and it became a widely used tool in pain studies. The aim of this study was to translate and culturally adapt the original English version of the CSQ into Turkish version and to assess the validity and reliability of this instrument in patients with chronic musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

* Being eighteen years old or older,
* being diagnosed with chronic musculoskeletal pain (at least 6 months),
* Being a native Turkish speaker and being able to read Turkish,
* Receiving no treatment between test-retest assessments.

Exclusion Criteria:

* Inability to complete the form due to significant psychiatric or psychological disorder,
* having a neurological disease,
* Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic musculoskeletal pain.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Reliability of Coping Strategies Questionnaire (CSQ) | 1 year
  As a result of the internal consistency analysis, Cronbach's Alpha coefficient was found to be 0.913. This value indicates that the scale has a high level of internal consistency.
  For the test-retest analysis of the Turkish version (CSQ-T), a 48-hour time interval was considered to be appropriate, and 40 participants were included in the test. As a result of the analysis, the ICC value was computed for the total score of the scale, which was found to be fairly high (0.876). The results revealed that both the sub-parameters and the total score of the CSQ, and thus the CSQ itself are stable over time.
  Based on these findings, the Turkish version of the questionnaire appears to have high reliability.
Validity of Coping Strategies Questionnaire (CSQ) | 1 year
  Construct validity was measured by comparing the responses of the scales of the CSQ-T with the responses of the scales of the HADS and SF-36. The total CSQ-T correlated to the anxiety subscale of the HADS with a score of r:-0.603 and to the depression subscale of the HADS with scores of r:-0.471. The SF-36 "PCS" (r: 0.790) and "MCS" (r:822) subscales were observed to have a good and very good correlation with the total score of CSQ-T.
  Based on these findings, the Turkish version of the questionnaire appears to have high validity.

CONTACTS AND LOCATIONS:
Overall Officials: Selda BAŞAR, Study Chair — Gazi University
Locations (1):
- Gazi University, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No